CLINICAL TRIAL: NCT01755585
Title: Irradiation Modulates the Pharmacokinetics of Anticancer Drugs
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH No. 099148-F
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Rectal Cancer; Cervical Cancer
Keywords: Radiation therapy; 5-fluorouracil; Cisplatin; Pharmacokinetics; Matrix Metalloproteinase
MeSH Terms: conditions — Rectal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood collection

GROUPS / COHORTS (2):
- C/T-RT group: Chemotherapy (C/T) is applied in the morning. After 2-4 hrs, radiotherapy (RT) is delivered (according to the clinical practice)
- RT-C/T group: Radiotherapy (RT) is delivered in the morning. After 2-4 hrs, chemotherapy (C/T) is applied (according to the clinical practice).

SUMMARY:
Radiation therapy (RT) is used as an effective local treatment modality to inhibit cell proliferation, induce cell death and suppress tumor growth. To improve the treatment outcome, in terms of both locoregional control and survival, the concurrent use of chemotherapy during radiation therapy (CCRT) is now the standard treatment for various malignancies, especially locally advanced cancers. Among the drugs used to enhance RT effect, 5-fluorouracil (5-FU) is one of the most commonly used chemotherapeutic agents of CCRT.

In the past, RT was solely used as a local treatment and its effect was estimated by local effect model. However, growing evidence shows that irradiation has direct DNA damage-dependent effects as well as sending signals to neighboring cells. Recently, we reported that abdominal irradiation could significantly modulate the systemic pharmacokinetics of 5-FU at 0.5 Gy, off-target area in clinical practice, and at 2 Gy, the daily treatment dose for target treatment in an experimental rat model. Additionally, the results from a clinical investigation showed that colorectal cancer patients with lower AUC of 5-FU during adjuvant chemotherapy had lower disease-free survival. Taken together, these lines of evidence support the importance and necessity to search for the mediators responsible for the unexpected effect of local RT on systemic pharmacokinetics of chemotherapeutic agents, such as 5-FU.

In the present study, the investigators investigated whether the phenomena and mechanism of RT-PK is a fact for different anticancer drugs in human.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) performance status of 0 or 1
* Age 18-80 years
* Locally advanced rectal cancer
* Locally advanced cervical cancer

Exclusion Criteria:

* Cancer history
* Abnormal liver and renal disease
* Immune disease
* Hematological disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chemotherapy-naive patients with histologically confirmed, locally advanced rectal adenocarcinoma and cervical cancer, who were prepared for concurrent chemoradiation therapy, were consecutively enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

REFERENCES:
- [Derived] Hsieh CH, Hou ML, Chiang MH, Tai HC, Tien HJ, Wang LY, Tsai TH, Chen YJ. Head and neck irradiation modulates pharmacokinetics of 5-fluorouracil and cisplatin. J Transl Med. 2013 Sep 26;11:231. doi: 10.1186/1479-5876-11-231. PMID 24066670